CLINICAL TRIAL: NCT05132088
Title: Efficacy and Safety of Oral Semaglutide 50 mg Once Daily in East Asian Participants With Overweight or Obesity
Brief Title: Research Study to Investigate How Well Semaglutide Tablets Taken Once Daily Work in East Asian People Who Are Overweight or Living With Obesity
Acronym: OASIS 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9932-4738; U1111-1258-7561 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- oral semaglutide 50 mg once daily (Experimental): All participants will get semaglutide or placebo tablets, 1 tablet every morning.
  Interventions: Drug: semaglutide 50 mg
- oral semaglutide placebo once daily (Placebo Comparator): All participants will get semaglutide or placebo tablets, 1 tablet every morning.
  Interventions: Drug: placebo (semaglutide)

INTERVENTIONS:
Drug: semaglutide 50 mg — Participants will have semaglutide for 68 weeks and will have 1 tablet every morning.
  Dose gradually increased to 50 mg.
  Arms: oral semaglutide 50 mg once daily
Drug: placebo (semaglutide) — Participants will have placebo tablets for 68 weeks and will have 1 tablet every morning.
  Arms: oral semaglutide placebo once daily

SUMMARY:
Novo Nordisk are doing this study to see if semaglutide tablets can be used as a treatment to help people living with overweight or obesity lose weight.

This study will look at the change in participants' body weight. Participants will either get semaglutide tablets (new medicine) or placebo tablets ('dummy' medicine that looks like semaglutide but has no effect on the body). For a fair comparison, people are divided into two groups at random by a computer. This process is called randomisation.

Semaglutide tablets are new medicine being tested to treat overweight and obesity. Doctors in many countries can already prescribe semaglutide tablets at lower doses to treat type 2 diabetes.

Participants will get semaglutide or placebo tablets for 68 weeks and will need to take 1 tablet every morning.

In addition to taking the medicine, participants will have talks with study staff about:

* healthy food choices
* how to be more physically active
* what participants can do to lose weight The study will last for about 1½ year. Participants will have 14 clinic visits and 7 phone calls with the study healthcare professional.

Blood samples will be taken at 12 visits. Women cannot take part if pregnant, breast-feeding or planning to get pregnant during the study period. If participants are a woman and are able to become pregnant, participants will be checked for pregnancy via urine tests.

ELIGIBILITY:
Inclusion criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Body mass index (BMI) of greater than or equal to 27.0 kg/m^2 with greater than or equal to 2 weight related comorbidities (treated or untreated) according to the JASSO guideline or BMI greater than or equal to 35.0 kg/m^2 with greater than or equal to1 weight related comorbidity (treated or untreated) according to the JASSO guideline. At least one comorbidity should be hypertension, dyslipidaemia or type 2 diabetes (T2D)
* History of at least one self-reported unsuccessful dietary effort to lose body weight

For participants with T2D at screening the following inclusion criteria apply in addition to criteria 1-4:

* Diagnosed with T2D greater than or equal to 180 days prior to screening
* Treated with either diet and exercise alone or stable treatment (same drug(s), dose and dosing frequency) for at least 60 days prior to the day of screening with up to 3 oral antidiabetic drugs (OADs) alone or in any combination (metformin, α-glucosidase (AGI), sulphonylureas (SU), glinides, SGLT2i (sodium-glucose co-transporter 2 inhibitor) or thiazolidinediones)
* HbA1c 7.0-10.0% (53-86 mmol/mol) (both inclusive) as measured by central laboratory at screening

Exclusion criteria:

Participants without T2D only:

* HbA1c greater than or equal to 6.5% (48 mmol/mol) as measured by the central laboratory at screening
* History of type 1 or type 2 diabetes
* Treatment with glucose-lowering agent(s) within 90 days prior to screening
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of eGFR brlow 15 ml/min/1.73 m^2 according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation as defined by kidney disease improving global outcomes (KDIGO) 2012 classification by the central laboratory at screening

Participants with T2D at screening only:

* Treatment with any medication for the indication of diabetes other than stated in the inclusion criteria within the past 60 days prior to screening
* Receipt of any other anti-diabetic investigational drug within 90 days prior to screening for this study, or receipt of any investigational drugs not affecting diabetes within 30 days prior to screening for this study
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed by an ophthalmologist or another suitably qualified health care provider within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Renal impairment measured as eGFR value of below 30 mL/min/1.73 m^2 according to CKD EPI creatinine equation as defined by KDIGO 2012 classification by the central laboratory at screening
* In participants treated with SGLT2i, renal impairment measured as eGFR value of below 60 mL/min/1.73 m^2 according to CKD EPI creatinine equation as defined by KDIGO 2012 classification by the central laboratory at screening

The following criteria apply to all participants:

Obesity-related:

* Treatment with any medication indicated for weight management within 90 days prior to screening
* Previous or planned (during the study period) obesity treatment with surgery or a weight loss device. However, the following are allowed: (1) liposuction and/or abdominoplasty, if performed greater than 1 year prior to screening, (2) lap banding, if the band has been removed greater than 1 year prior to screening, (3) intragastric balloon, if the balloon has been removed greater than 1 year prior to screening or (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed greater than 1 year prior to screening
* Uncontrolled thyroid disease per investigators discretion
* A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Percentage-point
Achievement of body weight reduction greater than or equal to 5% (Yes/No) | At end of treatment (week 68)
  Count of participants

SECONDARY OUTCOMES:
Achievement of body weight reduction greater than or equal to 10% (Yes/No) | At end of treatment (week 68)
  Count of participants
Change in Physical function domain (5-items) score (IWQOL-Lite-CT) | From baseline (week 0) to end of treatment (week 68)
  Score points
Achievement of body weight reduction greater than or equal to 15% (Yes/No) | At end of treatment (week 68)
  Count of participants
Achievement of body weight reduction greater than or equal to 20% (Yes/No) | At end of treatment (week 68)
  Count of participants
Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 68)
  Count of participants
Change in waist circumference measured according to the JASSO guideline | From baseline (week 0) to end of treatment (week 68)
  Messured in CM
Change in Visceral Fat Area (VFA) measured by CT scan in a subset of the Japanese study population | From baseline to end of treatment (week 68)
  %-point
Change in Visceral Fat Area (VFA) measured by CT scan in a subset of the Japanese study population | From baseline to end of treatment (week 68)
  Messured in cm^2
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 68)
  Messured in mmHg
Change in diastolic blood pressure | From randomisation (week 0) to end of treatment (week 68)
  Messured in mmHg
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 68)
  %-point
Change in lipids: Total cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: high density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: very-low density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: Triglycerides | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: Free fatty acids | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in high sensitivity C Reactive Protein | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Number of treatment emergent adverse events | From baseline (week 0) to end of study (week 75)
  Count of events
Number of serious adverse events | From baseline (week 0) to end of study (week 75)
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (13):
- Japan (9):
  - Iryouhoujinsyadan Shoureikan Shinsapporo Seiryou Hospital, Sapporo, Hokkaido
  - Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - OCROM Clinic, Suita-shi, Osaka
  - Naka Kinen Clinic, Ibaraki
  - Toranomon Hospital, Endocrinology and Metabolism, Minato-ku, Tokyo
  - Osaka University Hospital, Osaka
  - Takatsuki Red Cross Hospital, Osaka
  - Tokyo Center Clinic, Tokyo
  - ToCROM Clinic, Tokyo
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Kangbuk Samsung Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Kadowaki T, Heftdal LD, Ko HJ, Overvad M, Shimomura I, Thamattoor UK, Kim KK; OASIS 2 Investigators. Oral Semaglutide in an East Asian Population With Overweight or Obesity, With or Without Type 2 Diabetes: The OASIS 2 Randomized Clinical Trial. JAMA Intern Med. 2025 Oct 1;185(10):1206-1217. doi: 10.1001/jamainternmed.2025.3599. PMID 40758358